CLINICAL TRIAL: NCT05220501
Title: Optimization of Prostate Biopsy - Micro-Ultrasound Versus MRI: A 3-arm Randomized Controlled Trial Evaluating the Role of 29MHz Micro-ultrasound in Guiding Prostate Biopsy in Men With Clinical Suspicion of Prostate Cancer.
Brief Title: Optimization of Prostate Biopsy - Micro-Ultrasound Versus MRI
Acronym: OPTIMUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Exact Imaging (Industry)
Responsible Party: Principal Investigator, Dr. Laurence Klotz, Affiliate Scientist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EVU-2021-001
Record Dates: First submitted 2021-12-09; First posted 2022-02-02 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer
Keywords: prostate; prostate biopsy; micro-ultrasound
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: All three arms will be active at the same time and subjects will be randomized to one arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Microultrasonography only (Active Comparator): Subjects will undergo biopsy using micro-ultrasound only.
  Interventions: Diagnostic Test: Microultrasonography Targeted Biopsy
- Microultrasonography + MRI (Active Comparator): Subjects will undergo fusion biopsy using mpMRI and micro-ultrasound
  Interventions: Diagnostic Test: Microultrasonography Targeted Biopsy; Diagnostic Test: MRI Targeted Biopsy
- MRI + Conventional Ultrasonography (Active Comparator): Subjects will undergo biopsy using mpMRI fused with regular ultrasound
  Interventions: Diagnostic Test: MRI Targeted Biopsy

INTERVENTIONS:
Diagnostic Test: Microultrasonography Targeted Biopsy — All subjects will be biopsied no matter their arm randomization. In this group, MicroUS targets will be identified and sampled.
  Arms: Microultrasonography + MRI; Microultrasonography only
Diagnostic Test: MRI Targeted Biopsy — All subjects will be biopsied no matter their arm randomization. In this group, mpMRI targets will be identified and sampled.
  Arms: MRI + Conventional Ultrasonography; Microultrasonography + MRI

SUMMARY:
OPTIMUM is a study designed to compare the ability of ultra-high resolution transrectal micro-ultrasound (microUS) and multiparametric MRI (mpMRI)/US fusion to guide prostate biopsy.

DETAILED DESCRIPTION:
The purpose of the Clinical Investigation Plan and Study Protocol is to present information for the OPTIMUM clinical investigation, including the scientific basis for the study, the procedural details, the ExactVu High Resolution Micro-Ultrasound System, its safety details, and administrative details. It has been designed in such a way as to optimize the scientific validity and reproducibility of the results of the study in accordance with current clinical knowledge and practice so as to fulfill the objectives of the investigation.

ELIGIBILITY:
Inclusion Criteria:

* Men indicated for prostate biopsy due to elevated Prostate Specific Antigen and/or abnormal Digital Rectal Examination
* No history of prior prostate biopsy
* No history of genitourinary cancer, including prostate cancer
* 18 years or older
* No contraindications to biopsy
* No contraindications to mpMRI
* No history of mpMRI for clinical investigation of prostate cancer within 12 months prior to screening and enrollment in the study

Exclusion Criteria:

* History of prior prostate biopsy
* History of genitourinary cancer, including prostate cancer
* Contraindications to biopsy
* Contraindications to mpMRI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants need to have a prostate and have been referred to a urologist
Enrollment: 804 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Klotz, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (22):
- United States (5):
  - UCLA, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - University of Florida Health, Gainsville, Florida
  - Johns Hopkins, Baltimore, Maryland
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
- Ordensklinikum Elisabethinen, Linz, Austria
- Hopital Delta, Brussels, Belgium
- Canada (5):
  - University of Alberta, Edmonton, Alberta
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network - Princess Margaret Hospital, Toronto, Ontario
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Hôpital du Sacré-Cœur de Montréal, Montreal, Quebec
- France (2):
  - Centre Hospitàlier Martigues, Hôpitaux de Provence, Martigues
  - L'Institut Mutualiste Montsouris, Paris
- Germany (4):
  - University of Brandenburg, Brandenburg, Brandenburg
  - University of Magdeburg, Magdeburg, Saxony-Anholt
  - ProUro, Berlin
  - University of Tuebingen, Tübingen
- Humanitas, Milan, Italy
- Spain (3):
  - Urologica Clinica Bilbao, Bilbao
  - Madrid ROC, Madrid
  - ICUA Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No
Contractual limitations

REFERENCES:
- [Background] Kinnaird A, Luger F, Cash H, Ghai S, Urdaneta-Salegui LF, Pavlovich CP, Brito J, Shore ND, Struck JP, Schostak M, Harland N, Rodriguez-Socarras M, Brisbane WG, Lughezzani G, Toledano H, Ouertani MS, Macek P, Fung C, Tu W, Gusenleitner A, Gunzel K, Incze PF, George AK, Pereira JG, Jansen R, Renzulli J 2nd, Klotz L; OPTIMUM Investigators. Microultrasonography-Guided vs MRI-Guided Biopsy for Prostate Cancer Diagnosis: The OPTIMUM Randomized Clinical Trial. JAMA. 2025 May 20;333(19):1679-1687. doi: 10.1001/jama.2025.3579. PMID 40121537

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment opened Dec 2021. Study closed September 6, 2024 after interim analysis endpoints were met for primary outcome. 804 participants recruited, 802 patients randomized. 2 participants withdrew consent prior to randomization. 678 participants were biopsied from 20 centres (hospital and clinics).
Pre-assignment Details: Assignment done at point of enrollment
Groups:
- Microultrasonography: Participants received microultrasonography-guided targeted biopsy and systematic sampling
- Microultrasonography/MRI: Participants received microultrasonography/mpMRI-fusion guided targeted biopsy and systematic sampling
- MRI/conventional ultrasonography: Participants received mpMRI/conventional ultrasonography guided targeted biopsy and systematic sampling
Period: Overall Study
Arm/Group | Microultrasonography | Microultrasonography/MRI | MRI/conventional ultrasonography
Started | 137 | 263 | 402
Completed | 121 | 226 | 331
Not Completed | 16 | 37 | 71
Not completed — Withdrawal by Subject | 11 | 21 | 32
Not completed — Awaiting biopsy at time of interim analysis. Study closed. Primary endpoint met | 5 | 16 | 39

BASELINE CHARACTERISTICS:
Population: 678 participants were randomized and received intervention at the time of interim analysis and study close. 804 participants were enrolled, 2 withdrew prior to randomization leavin
Groups:
- Microultrasonography/MRI: Participants received microultrasonography/MRI-fusion guided targeted biopsy and systematic sampling
- MRI/Conventional Ultrasonography: Participants received MRI/conventional ultrasonography guided targeted biopsy and systematic sampling
- Total: Total of all reporting groups
Arm/Group | Microultrasonography | Microultrasonography/MRI | MRI/Conventional Ultrasonography | Total
Number analyzed (Participants) | 121 | 226 | 331 | 678
Age, Categorical [Count of Participants; unit: Participants] — Male participants greater than or equal to 18 years of age
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 55 | 100 | 161 | 316
    >=65 years | 66 | 126 | 170 | 362
Sex: Female, Male [Count of Participants; unit: Participants] — Study only applicable to those at risk for prostate cancer
  Participants
    Female | 0 | 0 | 0 | 0
    Male | 121 | 226 | 331 | 678
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African descent | 3 | 8 | 16 | 27
  Asian descent | 3 | 9 | 13 | 25
  Caucasian descent | 105 | 180 | 277 | 562
  Hispanic descent | 9 | 20 | 15 | 44
  Not stated/not reported | 1 | 9 | 10 | 20
PSA (Prostate Specific Antigen) [Median (Inter-Quartile Range); unit: ng/ml] — PSA (Prostate Specific Antigen) at time of enrollment
  ng/ml | 7.2 [5.5 to 11.0] | 7.0 [5.2 to 9.4] | 6.7 [5.1 to 9.5] | 6.8 [5.2 to 9.8]
Digital Rectal Exam (DRE) [Count of Participants; unit: Participants] — Count of participants where DRE was suspicous at the time of enrollment
  Participants | 25 | 48 | 81 | 154
Positive family history for prostate cancer [Count of Participants; unit: Participants] — Positive family history for prostate cancer at the time of enrollment
  Participants | 29 | 55 | 78 | 162

OUTCOME MEASURES:

1. Secondary Outcome: Difference in csPCa Rate Between MicroUS/MRI- Guided Fusion Biopsy and MRI/Conventional Ultrasonography Guided Fusion Biopsy
Description: The secondary outcome, detection of clinically significant prostate cancer by combined microultrasonography/mpMRI-guided fusion biopsy vs mpMRI/conventional ultrasonography-guided fusion biopsy.
Time Frame: Immediately after biopsy
Measure: Count of Participants; unit: Participants
Groups:
- Microultrasonography/MRI: MicroUS/mpMRI ultrasonography guided Biopsy with synchronous systematic biopsy
- MRI/ conventional ultrasonography: mpMRI/conventional ultrasonography guided Biopsy with synchronous systematic biopsy
Arm/Group | Microultrasonography/MRI | MRI/ conventional ultrasonography
Number analyzed (Participants) | 226 | 331
Participants | 106 | 141

2. Primary Outcome: Difference in Detection of Gleason Grade Group 2 or Higher Cancers Using Microultrasonography Plus Systematic Biopsy vs mpMRI/Conventional Ultrasonography Plus Systematic Biopsy
Description: As per protocol, the microultrasonography group for the primary outcome is defined as the microultrasonography-guided biopsy group and the blinded portion (microultrasound targets are identified prior to the unblinding of the MRI targets identified in the microultrasonography/mpMRI group).
  Difference in the detection rate of clinically significant prostate cancer (defined as equal to Gleason Grade Group 2 or higher) found using microultrasonography-guided biopsy, including targeted and systematic samples from the microultrasonography group and the mpMRI-blinded portion of the microultrasonography/mpMRI group, versus mpMRI/conventional ultrasonography-guided biopsy, including targeted and systematic samples from the mpMRI/conventional ultrasonography group.
Time Frame: Post biopsy
Population: As per protocol, the rate of clinically significant prostate cancer found, was compared between participants who underwent microultrasonography (57 of 121 from microultrasonography group and 103 of 226 from the MRI blinded portion of the microultrasonography/mpMRI group) from those participants who underwent mpMRI/conventional ultrasonography-guided biopsy.
Measure: Count of Participants; unit: Participants
Groups:
- Microultrasonography: Microultrasonography-guided biopsy, including targeted and systematic samples from the microultrasonography group and the mpMRI-blinded portion of the microultrasonography/mpMRI group
- MRI/Conventional ultrasonography: mpMRI/conventional ultrasonography-guided biopsy, including targeted and systematic samples from the mpMRI/conventional ultrasonography group
Arm/Group | Microultrasonography | MRI/Conventional ultrasonography
Number analyzed (Participants) | 347 | 331
Participants | 160 | 141
Statistical Analysis 1: Comparison: Microultrasonography vs MRI/Conventional ultrasonography; Test type: Non-Inferiority — The justification of the noninferiority margin is based on review of 11 studies reporting on the benefit of multiparametric MRI-directed biopsy over systematic biopsy. The differences between the multiparametric MRI-directed biopsy and systematic biopsy were tabulated and found to range from 5%to 18%. Panel selected 10% noninferiority and a 1-sided α of .025 as a reasonable threshold that would demonstrate clinically similar outcomes; p < 0.001, Jeffreys interval

ADVERSE EVENTS:
Time Frame: 7-days post biopsy
Groups:
- Microultrasonography/MRI: Participants received microultrasonography-guided targeted biopsy and systematic sampling
Arm/Group | Microultrasonography | Microultrasonography/MRI | MRI/conventional ultrasonography
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/226 | 0/331
Serious Adverse Events (participants affected / at risk) | 0/121 | 0/226 | 0/331
Other Adverse Events (participants affected / at risk) | 0/121 | 1/226 | 9/331
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microultrasonography (N=121) | Microultrasonography/MRI (N=226) | MRI/conventional ultrasonography (N=331)
Infection (Surgical and medical procedures) | 0 (0) | 0 (0) | 3 (3)
Urinary Tract Disorders (Renal and urinary disorders) | 0 (0) | 1 (1) | 5 (5) — Hematuria, Increase in LUTS (lower urinary tract symptoms) and urinary retention
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study mandated biopsy for all men in the trial. Currently, many men with PI-RAD 1 or 2 scores and favorable PSA density avoid biopsy. Trial design was open-label so no study member was blinded to biopsy technique. MRI/ultrasonography fusion device was not standardized across sites. Investigators used the device they were most comfortable with. Study restricted to biopsy naive men, therefore did not address microultrasonography in other clinical scenarios (i.e. active surveillance).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/01/NCT05220501/Prot_SAP_001.pdf